CLINICAL TRIAL: NCT03938597
Title: Investigation of Serious Adverse Events Following Vaccination Against Yellow Fever: Emphasis on Genetic Basis and Biological Markers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: ASCLIN002/2016
Record Dates: First submitted 2018-04-05; First posted 2019-05-06 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Drug-Related Side Effects and Adverse Reactions
Keywords: yellow fever vaccine; genetic factors; viscerotropic disease; neurological disease
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It concerns an investigation aiming to investigate genetic biological(s) marker(s) which allow to identify individuals who have risk of serious adverse events to the yellow fever vaccine. This testing is free of hypothesis, because these markers are still unknown. There is no intervention, and it is not possible to establish primary and secondary outcomes.

DETAILED DESCRIPTION:
The rational for the immunological study by LATIM is the observation made by the group that individuals vaccinated with the 17DD yellow fever vaccine show significant alterations on the levels of expression of genes such as CLEC5A, IFNG, IL6, RNASEL, IRF7, IRF9, STAT2 e OAS1 (8). The study which will be conducted by the Rockefeller University will be focused in the qualitative analysis of the genome and exome of volunteers. The study in LATIM will be focused in the quantitative analysis of mRNA, which, together with the results of sequencing, may help in the search for biomarkers. As the expression of mRNA is restricted to the acute phase of the adverse event, it will be done only during the first 30 days after the beginning of the adverse event.

ELIGIBILITY:
Inclusion criteria:

* Evidence of a systemic reaction in two or more organs within one month of vaccination with yellow fever vaccine;
* Laboratory evidence of yellow fever vaccine virus (at least one):

Positive culture for more than 7 days after vaccination; RT-PCR ≥ 3 log10 PFU/mL at any day after vaccination; Positive RT-PCR more than 14 days after vaccination; Presence of vaccine virus in tissue by culture, RT-PCR or immunohistochemistry.

* Laboratory exclusion of relevant differential diagnosis such as leptospirosis, viral hepatitis and arboviruses.
* Cases not obeying these strict criteria but that could be plausibly YEL-AVD or YEL-AND may be included, if approved by the investigator or co-investigators.

Exclusion Criteria:

* Cases with adverse event after yellow fever vaccine not severe.

Ages: 9 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will recruit cases of severe adverse event after yellow fever vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-01-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Genetic markers | Time frame: 5 years
  Whole exome sequencing (WES) will be performed in YEL-AVD cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Assessoria Clinica / Bio-Manguinhos / Fiocruz, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No